CLINICAL TRIAL: NCT06465862
Title: TruTag: Development of a Silica Microparticle Taggant System to Measure Antiretroviral Pharmacotherapy Adherence
Brief Title: Development of a Silica Microparticle Taggant System to Measure ART Adherence
Acronym: TruTag
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Trutag Technologies (Unknown); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Peter R Chai MD, Associate Professor of Emergency Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2024p001248
Record Dates: First submitted 2024-06-05; First posted 2024-06-20 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Hiv; Medication Adherence; Compliance, Medication
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Medication Adherence | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Intervention Model Description: Single arm pilot demonstration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TruTag System (Experimental): Participants will operate the TruTag system daily to record their adherence to TruTag-tagged Biktarvy for 90 days.
  Interventions: Device: TruTag System; Drug: Biktarvy Pill

INTERVENTIONS:
Device: TruTag System — TruTag technology system, consisting of microparticle-tagged Biktarvy and companion smartphone app.
Drug: Biktarvy Pill — Biktarvy prescribed with TruTag system and tagged with TruTag microparticles.

SUMMARY:
Developing technologies to help measure and provide tools to support medication-taking behaviors (medication adherence) is an important step to ending the human immunodeficiency virus (HIV) epidemic. TruTag Technologies has pioneered the use of a microparticle system that can be incorporated into the coating of medications may help users both identify the medication they are taking and record adherence events. By using a standard smartphone camera, shining light on TruTag-coated medications automatically identifies them to an onboard smartphone app which then indirectly records the adherence event. This study evaluates the real-world usability and feasibility of operating this system among people living with HIV (PLWH).

DETAILED DESCRIPTION:
This is an open-label pilot trial of N=15 PLWH who are prescribed Bictegravir/Emtricitabine/Tenofovir Alafenamide (Biktarvy) for antiretroviral therapy (ART). Participants will receive special TruTag-tagged Biktarvy and will be asked to scan their TruTag Biktarvy prior to ingesting it daily over 90 days. A companion smartphone app will record scans as an indirect measure of adherence. Included in the app will be a reminder system to nudge individuals to take their Biktarvy and a two-way text portal that allows participants to communicate securely with the study team. Participants will be screened and enrolled, and will then attend three monthly study visits, where the study team will assess adherence, dispense TruTag Biktarvy, and understand how the TruTag system is operated in the real world. At the final 90-day study visit, the study team will conduct a qualitative interview to explore acceptability and future design iterations of the TruTag system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older
2. Living with HIV
3. Currently prescribed and taking Biktarvy as ART for at least 3 months
4. Undetectable viral load in prior 6 months
5. Owns iPhone model 11 or higher (non-SE only)

Exclusion Criteria:

1. Not English-speaking
2. Unwilling to interact with the TruTag app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-15 (Estimated)

PRIMARY OUTCOMES:
Feasibility of TruTag to Measure Antiretroviral (ART) Adherence | 30, 60, 90 days
  Successful operation of the TruTag system will be measured over the 90-day study period. Total ingestions recorded by the TruTag system will be compared against total expected ingestions.
Acceptability of TruTag, via System Usability Scale | 90 days
  Acceptability will be measured via the System Usability Scale (SUS). The SUS is a 10-item measure of perceived usability of a technological system, scored on a 5-point Likert scale (1: strongly disagree, 5: strongly agree), with higher scores indicating greater perceived usability. A mean score of >68 will be used to indicate that the technology is acceptable.
Acceptability of TruTag, via Qualitative Interviews | 90 days
  Acceptability will be evaluated via qualitative interviews exploring participants' lived experiences operating the TruTag system and suggested improvements.

SECONDARY OUTCOMES:
Correlation of TruTag-Measured Adherence with Dried Blood Spot Concentrations | 90 days
  Preliminary accuracy of the TruTag system will be measured by correlating TruTag-detected ART adherence with tenofovir alafenamide concentrations in dried blood spots (DBS) collected at the 90-day visit.

CONTACTS AND LOCATIONS:
Overall Officials: Peter R Chai, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: No
Data available upon written communication with PI or study sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/62/NCT06465862/Prot_SAP_000.pdf